CLINICAL TRIAL: NCT02604329
Title: Feasibility Study of a Treatment Protocol of Pediatric Chemo- and Radiotherapy-induced Oral Mucositis by Low-level Laser Therapy
Brief Title: Feasibility Study of a Protocol to Treat Pediatric Oral Mucositis by Low-level Laser Therapy
Acronym: PEDIALASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/14/7421
Record Dates: First submitted 2015-10-20; First posted 2015-11-13 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-05

CONDITIONS: Oral Mucositis
Keywords: low level laser therapy; oral mucositis; child
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): Radiation : use of "Oncolase Digi" therapy laser diode
  Interventions: Device: "Oncolase Digi" therapy laser diode

INTERVENTIONS:
Device: "Oncolase Digi" therapy laser diode — The athermic phototherapy laser diode will be used by scanning the entire oral mucosa, including cheek and lip mucosa, gums, palate, tongue and floor of the mouth. It will be applied uniformly every two days as long as the grade of mucositis is 2 or more, with a fluence of 4J/cm², under two wavelengths (635 nm and 815 nm).
  * Cheeks will be scanned extra-orally with laser fiber during 50 seconds, at the fluence of 4J/cm², associating two wavelengths : infra-red (815 nm, 3850mW) and red (635 nm, 150mW).
  * Intra-orally, the fiber will be used to scan each area of mucositis during 30 seconds per area of 2 cm2, at 1cm from the mucosa; the power at 635 nm will be 150 milliwatts and 150 milliwatts at 815 nm.

SUMMARY:
Low Level Laser Therapy has been used for a few years in some pediatric hospital centers for chemo- and radiotherapy-induced oral mucositis care. It may promote ulceration's healing, limits mucositis severity and associated pain. As its use is recommended in the treatment of radio induced mucositis in adults, the level of evidence in pediatric studies does not allow a precise treatment protocol. The investigators present here the protocol of a feasibility study in the haemato-oncology department of the Children University Hospital of Toulouse, with the view to a future efficacy study.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of using low level laser therapy (LLLT) in the haemato-oncology department of the Children University Hospital of Toulouse. The feasibility will be considered as acceptable if 60% of patients hospitalized for oral mucositis had successfully benefit from the procedure. The secondary objectives are the evaluation of efficacy of LLLT on pain and mucositis grade, the evaluation of tolerance of this treatment and the medical time needed for this supportive care. The athermic phototherapy laser diode will be used by scanning the entire oral mucosa area. It will be applied uniformly every two days as long as grade of mucositis is 2 or more, with a fluence of 4J/cm², under two wavelengths (635 nm and 815 nm).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the oncology ward of the university hospital Toulouse France
* Onco-haematological paediatric patients treated by radio- and /or chemo-therapy, affected by an oral mucositis of WHO grade 2 to 4,
* lack of any physical or psychological disease which could interfere with the realization of the study.

Exclusion Criteria:

* Onco-haematological paediatric patients treated by radio- and /or chemo-therapy, affected by an oral mucositis of WHO's grade under 2
* Child suffering from epilepsy
* Patient wearing a cardiac pacemaker
* Patient not able to open their mouth at least 20 mm
* Patient refusing the wearing of safety goggles.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Success of the procedure for each included child | 7 days
  The procedure is successful when low level laser has been used on all the oral mucosa minimum 3 times in the first 7 days of mucositis of grade 2.
  The failure of the procedure is therefore declared if the laser was applied within 3 times within 7 days.
Participation rate | 1 year
  Number of included patients related to the number of patients hospitalized for mucositis with a WHO grade of 2 or more, in one year.

SECONDARY OUTCOMES:
Evaluation of mucositis grade | 7 days
  The World Health Organization (WHO) mucositis grade, before and after each laser application
Evaluation of the number of laser treatment sessions | 7 days
  Evaluation of the number of laser treatment sessions related to the mucositis episode
Pain evaluation with the HEDEN mucositis pain scale | 7 days
  Pain evaluation by medical caregivers with the HEDEN mucositis pain scale ("Hétero Evaluation Douleur Enfant")
Efficacy of low level laser therapy in the treatment of oral mucositis of grade 2 | 7 days
  Efficacy of low level laser therapy will be evaluate by medical caregivers with VAS (Visual Analogic Scale), before and after each laser application
Pain evaluation with the Venham scale | 7 days
  By medical caregiver delivering the laser treatment with the Venham scale modified by Veerkamp and OPS (Objective Pain Scale) for children under 6.
Evaluation of medical time needed for the treatment | 7 days
  Evaluation of the time spent with the patients for the treatment of oral mucositis by the medical staff

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle NOIRRIT-ESCLASSAN, PHD; DDS, Principal Investigator — Toulouse Children University Hospital
Locations (1):
- UH Toulouse, Toulouse, France

REFERENCES:
- [Result] Noirrit-Esclassan E, Valera MC, Vignes E, Munzer C, Bonal S, Daries M, Vaysse F, Puiseux C, Castex MP, Boulanger C, Pasquet M. Photobiomodulation with a combination of two wavelengths in the treatment of oral mucositis in children: The PEDIALASE feasibility study. Arch Pediatr. 2019 Jul;26(5):268-274. doi: 10.1016/j.arcped.2019.05.012. Epub 2019 Jul 4. PMID 31281038